CLINICAL TRIAL: NCT06509269
Title: Effect Of Intraoral Scanning Versus Desktop Scanning on The Retention Of Maxillary Denture Bases In Completely Edentulous Patients
Brief Title: Intraoral Scanning v.s Desktop Scanning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Ramy khalifa ashmawy, Ass.Lecturer, British University In Egypt
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Digital scanning
Record Dates: First submitted 2024-07-01; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Edentulous Jaw
Keywords: Intraoral Scanning; CAD/CAM denture; Desktop Scanning
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desktop Scanning (Active Comparator): Desktop scanning of Definitive Impression
  Interventions: Procedure: Desktop scanning
- IntraOral Scanning (Experimental): Intraoral scanning of edentulous Jaw
  Interventions: Procedure: intraoral scanning

INTERVENTIONS:
Procedure: intraoral scanning — Intraoral Scanning of edentulous Jaw
  Arms: IntraOral Scanning
Procedure: Desktop scanning — Desktop scanning of definitive impression
  Arms: Desktop Scanning

SUMMARY:
The aim of this study was to evaluate the effect of intraoral scanning versus desktop scanning on the retention and adaptation of maxillary denture bases in completely edentulous patients.

DETAILED DESCRIPTION:
The use of intra oral scanners (IOS) for rehabilitation of completely edentulous patients is still limited due to the difficulty in scanning large edentulous areas that are smooth and devoid of features. The stitching process can be defective, especially in the palatal area, where, the outmost deviations were reported in the palate when digitizing edentulous jaws with intraoral scanners. The main challenges for a fully digitized complete denture workflow are the digital impression of mobile tissues with functional border molding and the digital registration of the jaw relationship.

ELIGIBILITY:
Inclusion Criteria:

* Patients with well-developed ridge
* Firm healthy mucosa
* Free from any signs of inflammation

Exclusion Criteria:

* Patients having flabby ridge
* Decreased flow of saliva
* Limited mouth opening

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Retention of denture base | "through study completion, an average of 1 year"
  Measuring tool: Digital force meter, Measuring unit: Newton (N)
Adaptation of denture base | "through study completion, an average of 1 year"
  Measuring tool: Geomagic Control X software, Measuring Unit: Millimeter (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Ramy K Elashmawy, MSc, Principal Investigator — British University In Egypt
Locations (1):
- British University in Egypt, Cairo, Shorook, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osman RB, Alharbi NM. Influence of scan technology on the accuracy and speed of intraoral scanning systems for the edentulous maxilla: An in vitro study. J Prosthodont. 2023 Dec;32(9):821-828. doi: 10.1111/jopr.13633. Epub 2023 Jan 11. PMID 36571837
- [Background] Lo Russo L, Caradonna G, Troiano G, Salamini A, Guida L, Ciavarella D. Three-dimensional differences between intraoral scans and conventional impressions of edentulous jaws: A clinical study. J Prosthet Dent. 2020 Feb;123(2):264-268. doi: 10.1016/j.prosdent.2019.04.004. Epub 2019 May 29. PMID 31153614
- [Result] Manicone PF, De Angelis P, Rella E, Damis G, D'addona A. Patient preference and clinical working time between digital scanning and conventional impression making for implant-supported prostheses: A systematic review and meta-analysis. J Prosthet Dent. 2022 Oct;128(4):589-596. doi: 10.1016/j.prosdent.2020.11.042. Epub 2021 Mar 5. PMID 33678434